CLINICAL TRIAL: NCT01089257
Title: Subclinical Cardiovascular Impairments in Patients With Obstructive Sleep Apnea Syndrome
Brief Title: Cardiovascular Impairments and Obstructive Sleep Apnea Syndrome
Acronym: INFRASAS
Status: Terminated | Type: Observational
Why Stopped: Delayed inclusion at more than 14 years from the start of the study
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Centre Hospitalier Universitaire de Saint Etienne (Other); University Hospital, Clermont-Ferrand (Other); Hôpital de la Croix-Rousse (Other)
Responsible Party: Sponsor
Other Study IDs: 06PHR03
Record Dates: First submitted 2010-03-16; First posted 2010-03-18 (Estimated); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Subclinical Cardiovascular Impairments; Obstructive Sleep Apnea Syndrome
Keywords: Cardiovascular risks; Oxidative stress; Systemic inflammation; Endothelial function; Peripheral Arterial Tone; Positive Airway Pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Which are the anthropometric parameters and/or of severity of the syndrome of apnea of sleep (SAS) which make it possible to anticipate occurred of vascular anomalies, anatomical and/or functional precociously found among patients SAS? Secondary objectives:

1. Which are the anthropometric parameters and/or of severity of SAS allowing to anticipate occurred of early of the cardiac function and/or rhythmic anomalies found among patients SAS?
2. Do there exist biological markers who allow to anticipate the early vascular lesions or the anomalies beginners of the cardiac function?
3. Which are the cardiovascular effects of a treatment of SAS by Continuous Positive Pressure (PC) after 3 to 6 months of treatment?
4. Do the identified early cardiovascular attacks and/or the biological anomalies make it possible to predict occurred of cardiovascular events in this population of patients carrying SAS (followed longitudinal at 5 years)?

ELIGIBILITY:
Inclusion Criteria:

* Male or female from 18 to 78 years old
* Patients with obstructive sleep apnea syndrome (Apnea/Hypopnea index > 15)
* ambulatory patients
* patients who have signed the inform consent form
* patients with health insurance

Exclusion Criteria:

* Body Mass Index upper or equal to 30
* cardiovascular pathology except blood pressure hypertension
* known or treated diabetes
* pathologies with consequence on blood pressure regulation
* drugs intakes with consequence on blood pressure regulation
* patient with chronic obstructive pulmonary disease
* atrial fibrillation or more than 10/minute extrasystoles
* bedridden patients or patients with decreased mobility
* patients working at night or with shift work
* patients with carotid stenting or surgery history
* patients unable to sign the inform consent form
* patients already treated by cPAP or dental appliance for OSAS in the last 6 months
* pregnant or suckling female
* patients under supervision or trusteeship
* patients taking part in another clinical trial

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with obstructive sleep apnea syndrome (Apnea/Hypopnea index > 15)
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2021-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis JP PEPIN, ProfessorPhD, Principal Investigator — University Hospital, Grenoble
Locations (3):
- France (3):
  - France : Laboratoire d'explorations fonctionnelles du système nerveux - Functional explorations laboratory of nervous system, Clermont-Ferrand
  - France : Laboratoire EFCR - Functional cardiorespiratory explorations laboratory, Grenoble
  - France : Laboratoire EFCR - Functional cardiorespiratory explorations laboratory, Saint-Etienne

REFERENCES:
- [Background] Lattimore JD, Celermajer DS, Wilcox I. Obstructive sleep apnea and cardiovascular disease. J Am Coll Cardiol. 2003 May 7;41(9):1429-37. doi: 10.1016/s0735-1097(03)00184-0. PMID 12742277
- [Background] Parish JM, Somers VK. Obstructive sleep apnea and cardiovascular disease. Mayo Clin Proc. 2004 Aug;79(8):1036-46. doi: 10.4065/79.8.1036. PMID 15301332
- [Background] Shamsuzzaman AS, Gersh BJ, Somers VK. Obstructive sleep apnea: implications for cardiac and vascular disease. JAMA. 2003 Oct 8;290(14):1906-14. doi: 10.1001/jama.290.14.1906. PMID 14532320
- [Background] Marin JM, Carrizo SJ, Vicente E, Agusti AG. Long-term cardiovascular outcomes in men with obstructive sleep apnoea-hypopnoea with or without treatment with continuous positive airway pressure: an observational study. Lancet. 2005 Mar 19-25;365(9464):1046-53. doi: 10.1016/S0140-6736(05)71141-7. PMID 15781100
- [Background] Drager LF, Bortolotto LA, Lorenzi MC, Figueiredo AC, Krieger EM, Lorenzi-Filho G. Early signs of atherosclerosis in obstructive sleep apnea. Am J Respir Crit Care Med. 2005 Sep 1;172(5):613-8. doi: 10.1164/rccm.200503-340OC. Epub 2005 May 18. PMID 15901608
- [Result] Baguet JP, Boutin I, Barone-Rochette G, Levy P, Tamisier R, Pierre H, Boggetto-Graham L, Pepin JL. Hypertension diagnosis in obstructive sleep apnea: self or 24-hour ambulatory blood pressure monitoring? Int J Cardiol. 2013 Sep 1;167(5):2346-7. doi: 10.1016/j.ijcard.2012.11.037. Epub 2012 Nov 22. No abstract available. PMID 23176771
- [Derived] Stanke-Labesque F, Pepin JL, de Jouvencel T, Arnaud C, Baguet JP, Petri MH, Tamisier R, Jourdil JF, Levy P, Back M. Leukotriene B4 pathway activation and atherosclerosis in obstructive sleep apnea. J Lipid Res. 2012 Sep;53(9):1944-51. doi: 10.1194/jlr.P022814. Epub 2012 Jul 3. PMID 22761257